CLINICAL TRIAL: NCT00933491
Title: Risk Factors for Implant Bone Loss in Patients With Diabetes Mellitus: A Feasibility Cohort Study
Brief Title: Risk Factors for Implant Bone Loss in Patients With Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Tae-Ju Oh, Clinical Professor, University of Michigan
Other Study IDs: 2008-03
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Results first posted 2015-11-04 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes
Keywords: healthy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — saliva and plaque biofilm
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetic: Type II Diabetes
- Control: Non-diabetics

SUMMARY:
Dental implants are regarded as a standard of care in restoring missing teeth. Although there is a high prevalence of diabetics who receive dental implants, the relationship between dental implants and diabetes has not clearly been investigated.

A total of 32 subjects (14 patients with type II diabetes and 18 non-diabetes subjects) who have dental implants were recruited. The purposes of this research study were: (1) to evaluate diabetes patients to determine risk factors for bone loss at dental implants and teeth; and (2) to evaluate bone-resorptive biomarkers (proteins related to bone loss) present in saliva and blood serum, comparing the two groups.

DETAILED DESCRIPTION:
OBJECTIVE:

Regulators of peri-implant bone loss in patients with diabetes appear to involve multiple risk factors that have not been clearly elucidated. This study was conducted to explore putative local etiologic factors on implant bone loss in relation to type 2 diabetes mellitus, including clinical, microbial, salivary biomarker, and psychosocial factors.

MATERIALS AND METHODS:

Thirty-two subjects (divided into type 2 diabetes mellitus and non-diabetic controls), having at least one functional implant and six teeth, were enrolled in a 1-year longitudinal investigation. Analyses of clinical measurements and standardized intra-oral radiographs, saliva and serum biomarkers (via protein arrays for 20 selected markers), and plaque biofilm (via qPCR for eight periodontal pathogens) were performed at baseline and 1 year. In addition, the subjects were asked to respond to questionnaires to assess behavioral and psychosocial variables.

ELIGIBILITY:
Inclusion Criteria:

* be at least 40 years old
* have at least one dental implant that has been in function for at least 6 months
* have at least 6 natural teeth
* have good general oral health
* not be pregnant or breastfeeding or planning to become pregnant within the next year
* if you are a pre-menopausal woman you or your male partner must be surgically sterile or you must be using reliable birth control (i.e., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch) now and throughout the study or abstain from sex throughout the study

Exclusion Criteria:

* not have an active oral infection, including periodontitis and rampant caries
* not have a history of chronic systemic illness or infection, history of oral cancer, life expectancy of less than 5 years
* not have had cancer treatment in the last 12 months

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Type II diabetics and non diabetics with dental implants
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2008-11; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Ju Oh, DDS, MS, Principal Investigator — University of Michigan
Locations (1):
- Michigan Center for Oral Health Research, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Tatarakis N, Kinney JS, Inglehart M, Braun TM, Shelburne C, Lang NP, Giannobile WV, Oh TJ. Clinical, microbiological, and salivary biomarker profiles of dental implant patients with type 2 diabetes. Clin Oral Implants Res. 2014 Jul;25(7):803-12. doi: 10.1111/clr.12139. Epub 2013 Feb 27. PMID 23445216

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diabetic | Control
Started | 14 | 18
Completed | 14 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diabetic | Control | Total
Number analyzed (Participants) | 14 | 18 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 18 | 32
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 65 [51 to 80] | 64 [48 to 75] | 64.5 [48 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  United States | 14 | 18 | 32

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Bone Level
Description: Mean radiographic bone level at 12 months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diabetic | Control
Number analyzed (Participants) | 14 | 18
mm | 2.69 (.17) | 2.54 (.15)

2. Primary Outcome: Radiographic Bone Level
Description: Mean radiographic bone level at baseline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diabetic | Control
Number analyzed (Participants) | 14 | 18
mm | 2.59 (.15) | 2.71 (.14)

ADVERSE EVENTS:
Time Frame: 2 years
Description: We monitored for adverse events from subject recruitment phase to completion of the study which took two years (2008-2010).
Arm/Group | Diabetic | Control
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/18
Other Adverse Events (participants affected / at risk) | 0/14 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No